CLINICAL TRIAL: NCT03526120
Title: Acute Satiety and Energy Compensation After Consumption of a Pistachio Snack and Longer Term Consequences on Satiety, Anthropometry, and Body Composition After a Nutritional Intervention With Daily Consumption of the Pistachio Snack
Brief Title: Pistachio Intake, Satiety and Body Weight Control in Healthy Adult Women
Acronym: APIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rene' Yamashiro (Other)
Responsible Party: Sponsor-Investigator, Rene' Yamashiro, Sponsor-Investigator, American Pistachio Growers
Organization: American Pistachio Growers (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APIS; ID RCB : 20107-A031 (Registry Identifier: Agence Nationale de Sécurité du Médicament (ANSM, France)); APG01-0117 (Other: CreaBio-RA)
Record Dates: First submitted 2018-04-22; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Human subjects; Pistachio snack; Body mass index; Energy intake; Fat mass

STUDY DESIGN:
Intervention Model Description: Two parallel groups according a block randomization stratified on habitual energy intake and initial body weight (as in http://www.consort-statement.org/checklists/view/32--consort-2010/87-randomisation-type, § 8B). Randomisation: type).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pistachio diet (Experimental): Incorporates 44 g (1 serving) of pistachios into a daily diet
  Interventions: Other: Pistachio
- Control (No Intervention): No pistachio consumption

INTERVENTIONS:
Other: Pistachio — Dailly 44 g unsalted pistachios snack for 12 weeks
  Arms: Pistachio diet

SUMMARY:
The main goal of the study is to confirm that, due to their rich nutritional content in protein, polyunsaturated fatty acids, vitamins and minerals of interest (calcium and magnesium), the regular consumption of the recommended amount of pistachios by adult women will elicit appropriate satiety and compensation in the daily energy intake, and improve diet quality, anthropometry and body composition.

DETAILED DESCRIPTION:
The expected endpoint is to demonstrate that the daily consumption of a snack of pistachios by healthy women, as recommended in the next National Program for Nutrition and Health (program PNNS, France), elicits adequate satiety and does not induce weight gain but rather improves diet quality, body composition and body fat mass distribution (less abdominal fat).

The study will be a 16 weeks randomized controlled open trial, single-center, including two parallel groups of 30 female participants (block randomization stratified on habitual energy intake and initial body weight according to the consort-statement checklist).

The main working hypothesis is a demonstration of the "non inferiority" of the effects of the pistachio intervention on body weight versus no snack consumption. The investigators hypothesize that there will be no significant difference in body weight change due to pistachios consumption. The two-sided 95% confidence interval on the intra-patient difference (before minus after the pistachio intervention) will be provided through the appropriate contrasts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women;
2. Age: lower age limit 18 years, upper age limit: 50 years (included);
3. Body Mass Index: lower limit 19 kg/m²; upper limit 29.9 kg/m²; weight stable within ± 2 kg in the last 3 months;
4. Habitual energy intake, as indicated by an initial intake report (diary method, three days) within the 95% confidence interval (CI) of the habitual energy intake of a similar population (as provided by internal reference data collected by CREABio-RA from previous studies in similar conditions);
5. Participant not pregnant, not presently breast feeding or having breastfed in the last 3 months, and not planning to become pregnant during the study (negative pregnancy test at inclusion or morning of V1);
6. Pre-menopausal participant on effective contraception since at least 3 months (regular 28-day cycle) and who agree to continue their contraception throughout the study;
7. Participant registered with the French Social Security;
8. participant having signed informed consent

Exclusion Criteria:

1. Subject under legal protection or deprived of liberty by judicial or administrative decision.
2. Currently diagnosed somatic pathology;
3. On medication affecting metabolism, weight, energy intake, or energy expenditure in the last 6 months;
4. Major psychiatric disorder, particularly eating disorders as defined by the DSM-V;
5. High level of "Restrained Eating" or "Disinhibition", as revealed by the TFEQ or similar questionnaire;
6. Strong initial dislike of nuts, specially pistachios, as revealed by questioning about food habits initial dietary questionnaire;
7. Habitual consumption of pistachios as revealed by the 3-d intake report (more than twice a week);
8. Participants smoking more than 10 cigarettes per day or planning to stop smoking in the next 3 months;
9. Currently pregnant, lactating (as specified in article L1121-5 of the Public Health Code) or less than 6 month post-partum;
10. Any kind of food allergy, especially allergies or intolerance to nuts;
11. Participant not capable of understanding the constraints of the study, who does not agree to abide, and/or unable to communicate normally with investigators;
12. Person currently participating in another clinical study, or having used up her annual entitlement to compensation for participation in biomedical studies (4500 €).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  Body weight in kg

SECONDARY OUTCOMES:
Total daily energy intake | 12 weeks
  Total daily energy intake in kcal
Appetite ratings | 12 weeks
  Appetite ratings measured on visual analogic scalls of 100 mm
Body weight index | 12 weeks
  Body weight index in kg/m2
Body fat mass | 12 weeks
  Body fat mass in kg

CONTACTS AND LOCATIONS:
Overall Officials: Marc FANTINO, MD, PhD, Pr., Principal Investigator — CreaBio Rhône-Alpes
Locations (1):
- CreaBio Rhône-Alpes, Givors, Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fantino M, Bichard C, Mistretta F, Bellisle F. Daily consumption of pistachios over 12 weeks improves dietary profile without increasing body weight in healthy women: A randomized controlled intervention. Appetite. 2020 Jan 1;144:104483. doi: 10.1016/j.appet.2019.104483. Epub 2019 Oct 8. PMID 31604062